CLINICAL TRIAL: NCT03856515
Title: Gender Differences in Standardized Research E-Cigarette (SREC) Product Use, Acceptability, Reinforcement, and Nicotine Dependence Symptoms
Brief Title: Gender Differences in Switching From Smoking Regular Cigarettes to E-Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-0794; NCI-2018-03354 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0794 (Other: M D Anderson Cancer Center); U01DA047875 (NIH)
Record Dates: First submitted 2019-01-23; First posted 2019-02-27 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- E-Cig placebo dose followed by E-Cig nicotine dose (Experimental): Participants will be instructed to smoke their usual brand cigarette as they normally would in weeks 1-2 (Phase I) and to use only the SREC (with or without nicotine) in weeks 3-4 (Phase II) and in weeks 5-6 (Phase III). Participant assignment to SREC type at Phases II and III will be counter-balanced within group, with half of men and women receiving the placebo SREC during Phase II and half during Phase III. Participants will attend 4 laboratory visits with study investigators for 3 hours each over 6 weeks of study participation.
  Interventions: Drug: Nicotine Replacement; Other: Questionnaire Administration; Device: Electronic Cigarette
- E-Cig nicotine dose followed by E-Cig placebo dose (Experimental): Participants will be instructed to smoke their usual brand cigarette as they normally would in weeks 1-2 (Phase I) and to use only the SREC (with or without nicotine) in weeks 3-4 (Phase II) and in weeks 5-6 (Phase III). Participant assignment to SREC type at Phases II and III will be counter-balanced within group, with half of men and women receiving the placebo SREC during Phase II and half during Phase III. Participants will attend 4 laboratory visits with study investigators for 3 hours each over 6 weeks of study participation.
  Interventions: Drug: Nicotine Replacement; Other: Questionnaire Administration; Device: Electronic Cigarette

INTERVENTIONS:
Drug: Nicotine Replacement — Received NRT (Electronic Cigarette - With Nicotine)
  Other Names: Nicotine Replacement Therapy; NRT
Other: Questionnaire Administration — Ancillary studies
Device: Electronic Cigarette — Electronic Cigarette - with Nicotine
Device: Electronic Cigarette — Electronic Cigarette -without Nicotine

SUMMARY:
This early phase I trial studies potential differences between men and women when switching from the use of combustible cigarettes to the National Institute on Drug Abuse's Standard Research E-Cigarette (SREC). Studying the differences between men and women may increase understanding about the effects of switching from smoking regular cigarettes to electronic cigarettes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the effects of switching to nicotine versus (vs.) placebo standard research E-cigarettes (SRECs) from combustible cigarettes (CCs) on product use, product acceptability, reinforcement, and nicotine dependence symptoms among adult daily CC smokers.

II. To characterize the differences between male and female CC smokers when switching to nicotine versus (vs.) placebo SRECs from CCs on product use, product acceptability, reinforcement, and nicotine dependence symptoms.

EXPLORATORY OBJECTIVE:

I. To characterize which factors moderate or mediate the effects of switching to nicotine and placebo SRECs from CCs among male and female CC smokers.

OUTLINE:

Participants will be instructed to smoke their usual brand cigarette as they normally would in weeks 1-2 (Phase I) and to use only the SREC (with or without nicotine) in weeks 3-4 (Phase II) and in weeks 5-6 (Phase III). Participant assignment to SREC type at Phases II and III will be counter-balanced within group, with half of men and women receiving the placebo SREC during Phase II and half during Phase III. Participants will attend 4 laboratory visits with study investigators for 3 hours each over 6 weeks of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older
* Reports being a daily or non-daily smoker (any self-reported smoking in the past 30 days)
* Have an address where he/she can receive mail
* Able to follow verbal and written instructions in English and complete all aspects of the study as determined by PI
* Willing to have urine biospecimen samples taken, either in-home and returning them by mail, or in-person at an approved collection site.
* Willing to use tobacco-flavored study electronic cigarettes
* Agrees to comply with all MD Anderson institutional policies related to COVID-19 screening prior to any in-person research visit.
* The individual agrees to not engage in study procedures or interactions with study personnel while operating a vehicle.

Exclusion Criteria:

* Individuals who report depressive symptoms in the moderately severe or severe range on the PHQ-9 (scores of 15 or above) or who report current suicidal ideation on the PHQ-9
* Uncontrolled or unstable medical condition (e.g., uncontrolled hypertension, angina, diabetes).
* Evidence of cognitive deficits or instability that would preclude reliable study participation.
* Being pregnant, engaging in breast-feeding, or being of childbearing potential and engaging in sexual activity that could lead to pregnancy and is not protected by a medically acceptable, effective method of birth control while enrolled in the study, as determined by self-report. Medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD). Contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use.
* Considered by the investigator to be an unsuitable or unstable candidate (including but not limited to the following situation: unwilling or unable to comply with study procedures)
* Individuals who reside in an area that is outside of our shipping company's area of operation or in a jurisdiction outside of our medical staff's licensure (if unable to attend in-person clinic visits) AND who decline or are unable to come in to clinic to provide necessary samples and/or collect study products.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2026-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robinson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Robinson JD, Cui Y, Karam-Hage M, Blalock JA, Shete S, Kypriotakis G, Yang P, Cinciripini PM. Standardized research electronic cigarette acceptability among adult men and women who smoke combustible cigarettes. Psychol Addict Behav. 2025 Dec;39(8):780-791. doi: 10.1037/adb0001100. Epub 2025 Oct 6. PMID 41051837
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were adult individuals residing in the state of Texas who completed the study remotely.
Pre-assignment Details: Of the 1363 potential participants who responded to study advertising, 702 were screened for interest and eligibility. Of those screened, 130 were ineligible and 402 declined to participate. A total of 169 participants were randomized.
Groups:
- Phase 1: Usual Brand Cigarette Phase (Men): Two weeks (Phase 1; weeks 1-2) of smoking usual brand cigarettes (men)
- Phase 1: Usual Brand Cigarette Phase (Women): Two weeks (Phase 1; weeks 1-2) of smoking usual brand cigarettes (women)
- Phase 2 Placebo, Then Phase 3 Standardized Research Electronic Cigarette (SREC) (Men): Two weeks (Phase 2; weeks 3-4) of placebo Standardized Research Electronic Cigarette use, followed by two weeks (Phase 3; weeks 5-6) of nicotine Standardized Research Electronic Cigarette use (Men)
- Phase 2 Placebo, Then Phase 3 SREC (Women): Two weeks (Phase 2; weeks 3-4) of placebo Standardized Research Electronic Cigarette use, followed by two weeks (Phase 3; weeks 5-6) of nicotine Standardized Research Electronic Cigarette use (Women)
- Phase 2 SREC, Then Phase 3 Placebo (Men): Two weeks (Phase 2; weeks 3-4) of nicotine Standardized Research Electronic Cigarette use, followed by two weeks (Phase 3; weeks 5-6) of placebo Standardized Research Electronic Cigarette use (Men)
- Phase 2 SREC, Then Phase 3 Placebo (Women): Two weeks (Phase 2; weeks 3-4) of nicotine Standardized Research Electronic Cigarette use, followed by two weeks (Phase 3; weeks 5-6) of placebo Standardized Research Electronic Cigarette use (Women)
Period: Phase 1: Week 1-2
Arm/Group | Phase 1: Usual Brand Cigarette Phase (Men) | Phase 1: Usual Brand Cigarette Phase (Women) | Phase 2 Placebo, Then Phase 3 Standardized Research Electronic Cigarette (SREC) (Men) | Phase 2 Placebo, Then Phase 3 SREC (Women) | Phase 2 SREC, Then Phase 3 Placebo (Men) | Phase 2 SREC, Then Phase 3 Placebo (Women)
Started | 87 | 82 | 0 | 0 | 0 | 0
Completed | 87 | 82 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: Week 3-4
Arm/Group | Phase 1: Usual Brand Cigarette Phase (Men) | Phase 1: Usual Brand Cigarette Phase (Women) | Phase 2 Placebo, Then Phase 3 Standardized Research Electronic Cigarette (SREC) (Men) | Phase 2 Placebo, Then Phase 3 SREC (Women) | Phase 2 SREC, Then Phase 3 Placebo (Men) | Phase 2 SREC, Then Phase 3 Placebo (Women)
Started | 0 | 0 | 45 | 41 | 42 | 41
Completed | 0 | 0 | 39 | 38 | 40 | 35
Not Completed | 0 | 0 | 6 | 3 | 2 | 6
Period: Phase 3: Week 5-6
Arm/Group | Phase 1: Usual Brand Cigarette Phase (Men) | Phase 1: Usual Brand Cigarette Phase (Women) | Phase 2 Placebo, Then Phase 3 Standardized Research Electronic Cigarette (SREC) (Men) | Phase 2 Placebo, Then Phase 3 SREC (Women) | Phase 2 SREC, Then Phase 3 Placebo (Men) | Phase 2 SREC, Then Phase 3 Placebo (Women)
Started | 0 | 0 | 45 | 41 | 42 | 41
Completed | 0 | 0 | 36 | 37 | 38 | 32
Not Completed | 0 | 0 | 9 | 4 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Usual Brand Cigarette Phase (Men); Phase 1: Usual Brand Cigarette Phase (Women): Two weeks of smoking usual brand cigarettes followed by two weeks of using the Placebo (0% nicotine content) Standardized Research Electronic Cigarette (SREC) and the two weeks of using the Nicotine (5% nicotine content) SREC, with SREC order counterbalanced.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Usual Brand Cigarette Phase (Men) | Phase 1: Usual Brand Cigarette Phase (Women) | Total
Number analyzed (Participants) | 87 | 82 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.51 (11.26) | 44.57 (10.14) | 44.54 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 82 | 82
  Male | 87 | 0 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 7 | 22
  Not Hispanic or Latino | 72 | 75 | 147
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 23 | 44
  White | 47 | 55 | 102
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 10 | 0 | 10
Region of Enrollment [Number; unit: participants]
  United States | 87 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Day
Description: Mean cigarettes per day (CPD) smoked during the phase
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Cigarettes per Day
Groups:
- Usual Brand Cigarette Phase (Men): Two weeks of smoking usual brand cigarettes (Men)
- Placebo Standardized Research Electronic Cigarette Phase (Men): Two weeks of using the Placebo (0% nicotine content) Standardized Research Electronic Cigarette (Men)
- Nicotine Standardized Research Electronic Cigarette Phase (Men): Two weeks of using the Nicotine (5% nicotine content) Standardized Research Electronic Cigarette (Men)
- Usual Brand Cigarette Phase (Women): Two weeks of smoking usual brand cigarettes (Women)
- Placebo Standardized Research Electronic Cigarette Phase (Women): Two weeks of using the Placebo (0% nicotine content) Standardized Research Electronic Cigarette (Women)
- Nicotine Standardized Research Electronic Cigarette Phase (Women): Two weeks of using the Nicotine (5% nicotine content) Standardized Research Electronic Cigarette (Women)
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 83 | 81 | 82 | 76 | 79
Cigarettes per Day | 14.20 (9.01) | 4.08 (6.31) | 4.55 (7.25) | 14.09 (7.66) | 3.85 (5.30) | 3.63 (4.72)

2. Secondary Outcome: Electronic Cigarette Sessions Per Day
Description: Study electronic cigarette use measured by the mean number of sessions per day during each phase for male and female participants.
Time Frame: 2 weeks
Population: Electronic cigarette sessions per day were not assessed during the Usual Brand Cigarette phase.
Measure: Mean (Standard Deviation); unit: Sessions per day
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 0 | 83 | 81 | 0 | 76 | 79
Sessions per day |  | 11.32 (9.49) | 10.33 (8.93) |  | 10.78 (9.28) | 10.84 (10.84)

3. Secondary Outcome: Total Nicotine Equivalents (TNE)
Description: A measure of nicotine exposure, calculated as the sum of total nicotine, cotinine, 3'-hydroxycotinine, and nicotine N-oxide excreted in urine, collected at the end of each phase for male and female participants.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 73 | 73 | 77 | 66 | 69
ng/mL | 42.01 (37.40) | 30.98 (30.12) | 39.97 (36.44) | 41.19 (33.44) | 39.46 (38.80) | 41.75 (42.11)

4. Secondary Outcome: Anabasine
Description: A tobacco minor alkaloid (MA) excreted in urine collected at the end of each phase for male and female participants to evaluate nicotine product exposure.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 73 | 73 | 77 | 66 | 69
ng/mL | 92.69 (155.35) | 56.60 (97.03) | 71.45 (98.16) | 76.19 (92.95) | 72.90 (107.13) | 65.61 (83.24)

5. Secondary Outcome: Nicotelline
Description: as for outcome 4
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 73 | 73 | 77 | 66 | 69
ng/mL | 0.64 (4.53) | 0.38 (2.05) | 0.42 (2.92) | 1.63 (7.98) | 2.22 (8.42) | 1.08 (3.73)

6. Secondary Outcome: Perceived Health Risk Questionnaire (PHRQ)
Description: Evaluation of participants' beliefs about their risks of developing health conditions from cigarettes or electronic cigarette collected at the end of each phase for male and female participants. Range 1-10, with higher values indicating greater perceived risk of negative health outcomes.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 82 | 76 | 81 | 71 | 75
Units on a scale | 8.15 (2.18) | 8.35 (2.22) | 8.43 (2.06) | 9.05 (1.99) | 9.21 (1.79) | 9.23 (2.03)

7. Secondary Outcome: Product Evaluation Scales (PES)
Description: Evaluation of explicit cigarette or electronic cigarette product liking collected at the end of each phase for male and female participants. Range 1-7, with higher values indicating more unpleasant ratings.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 78 | 67 | 81 | 67 | 69
Units on a scale | 4.33 (0.98) | 3.30 (0.98) | 3.44 (1.04) | 4.51 (1.12) | 3.42 (1.17) | 3.73 (1.35)

8. Secondary Outcome: Implicit Association Test (IAT)
Description: Evaluation of implicit cigarette or electronic cigarette liking collected at the end of each phase for male and female participants. Range: -1 to 1, with more negative values indicating a more negative attitude toward the cigarette product
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 86 | 79 | 69 | 76 | 65 | 71
Units on a scale | -0.29 (0.53) | -0.17 (0.48) | -0.08 (0.50) | -0.32 (0.62) | -0.15 (0.40) | -0.25 (0.49)

9. Secondary Outcome: Brief Smoking Consequences Questionnaire-Adult (BSCQ-A)
Description: Evaluation of the perceived outcomes of cigarette or electronic cigarette use collected at the end of each phase for male and female participants. Range 0 to 9, with larger values indicating greater perceived negative consequences of cigarette use
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 82 | 76 | 81 | 71 | 75
Units on a scale | 4.56 (1.22) | 3.68 (1.25) | 3.54 (1.34) | 4.61 (1.25) | 3.70 (1.70) | 3.72 (1.84)

10. Secondary Outcome: Purchase Task Breakpoint Measure
Description: Evaluation of the Purchase Task Breakpoint measure (first price at which consumption goes to zero, i.e., unwilling to pay) for cigarettes or electronic cigarettes collected at the end of each phase for male and female participants. Range: 0.05 - 251, dollars per cigarette or per electronic cigarette puff with higher values indicating the willingness to smoke/vape at a higher price.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: $/cigarette or $/e-cigarette puff
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 64 | 61 | 76 | 53 | 59
$/cigarette or $/e-cigarette puff | 13.67 (22.12) | 7.06 (16.97) | 4.65 (9.69) | 14.25 (33.22) | 5.73 (10.64) | 7.44 (16.92)

11. Secondary Outcome: Purchase Task Demand Intensity Measure
Description: Evaluation of the Purchase Task Demand Intensity measure (consumption at the lowest price) for cigarettes or electronic cigarettes collected at the end of each phase for male and female participants. Range: 1 - 351, the number of cigarettes or electronic cigarette puffs with higher values indicating an intension to smoke/vape more when the price is set as 0
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: # of cigarettes or e-cigarette puffs
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 64 | 61 | 77 | 53 | 59
# of cigarettes or e-cigarette puffs | 20.52 (14.37) | 70.05 (69.59) | 59.08 (51.94) | 19.05 (13.14) | 48.06 (43.06) | 60.39 (56.06)

12. Secondary Outcome: Purchase Task Omax Measure
Description: Evaluation of the Purchase Task Omax measure (maximum financial expenditure on the product) for cigarettes or electronic cigarettes collected at the end of each phase for male and female participants. Range: 0.03 - 1001, the maximum expenditure in dollars on cigarettes or electronic cigarette puffs with higher values indicating greater expenditure
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: max spent $ on cigarettes or e-cig puffs
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 64 | 61 | 77 | 53 | 59
max spent $ on cigarettes or e-cig puffs | 17.96 (22.51) | 24.74 (72.92) | 11.73 (13.09) | 35.40 (127.18) | 13.51 (23.20) | 19.94 (65.14)

13. Secondary Outcome: Purchase Task Pmax Measure
Description: Evaluation of the Purchase Task Pmax measure (price at which expenditure is maximized) for cigarettes or electronic cigarettes collected at the end of each phase for male and female participants. Range: 0.01 - 1001, the price of the cigarette or electronic cigarette puffs when the Omax is reached
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: US Dollars per cigarette or per electron
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 64 | 61 | 77 | 53 | 59
US Dollars per cigarette or per electron | 4.64 (7.82) | 2.86 (7.97) | 1.65 (3.53) | 17.93 (114.14) | 2.36 (5.01) | 3.39 (8.39)

14. Secondary Outcome: Purchase Task Elasticity of Demand Measure
Description: Evaluation of the Purchase Task Elasticity of Demand measure (sensitivity of product consumption to increases in cost) for cigarettes or electronic cigarettes collected at the end of each phase for male and female participants. Range: 0.0001 - 2.69, the elasticity of the demand for cigarettes or electronic cigarette puffs, with higher values indicating a greater sensitivity in reducing the consumption in response to the price increases
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: % change quantity/% change price
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 82 | 64 | 61 | 77 | 53 | 59
% change quantity/% change price | 0.0070 (0.0040) | 0.0130 (0.0057) | 0.0177 (0.0068) | 0.008 (0.0040) | 0.026 (0.009) | 0.0298 (0.009)

15. Secondary Outcome: Fagerström Test for Cigarette Dependence (FTCD)
Description: Evaluation of cigarette dependence collected at the end of each phase for male and female participants. Range 0 to 10, with higher values indicating greater cigarette dependence
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 82 | 76 | 81 | 71 | 74
Units on a scale | 4.54 (2.09) | 3.71 (2.05) | 3.67 (2.07) | 4.7 (2.02) | 3.97 (2.28) | 3.88 (1.85)

16. Secondary Outcome: Penn State Electronic Cigarette Dependence Index (PSECDI)
Description: Evaluation of electronic cigarette dependence collected at the end of each phase for male and female participants. Range 0 to 20, with higher scores indicating greater electronic cigarette dependence
Time Frame: 2 weeks
Population: The PSECDI questionnaire was not administered during the Usual Brand Cigarette phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 0 | 78 | 67 | 0 | 67 | 69
Units on a scale |  | 7.78 (4.08) | 7.75 (3.97) |  | 8.87 (4.32) | 8.99 (4.36)

17. Secondary Outcome: Minnesota Nicotine Withdrawal Scale-Revised (MNWS)
Description: Evaluation of nicotine withdrawal symptoms collected at the end of each phase for male and female participants. Range 0 to 60, with higher scores indicating greater nicotine withdrawal
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 82 | 76 | 81 | 71 | 75
Units on a scale | 27.01 (7.98) | 27.02 (7.99) | 26.04 (7.62) | 28.81 (9.09) | 29.77 (9.77) | 28.08 (7.99)

18. Secondary Outcome: Questionnaire of Smoking Urges-Brief (QSU-Brief)
Description: Evaluation of the craving to smoke cigarettes collected at the end of each phase for male and female participants. Range 1 to 10, with higher values indicating greater urge to smoke
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 82 | 76 | 81 | 71 | 75
Units on a scale | 4.16 (2.57) | 3.35 (2.71) | 3.26 (2.83) | 4.25 (2.92) | 3.43 (3.04) | 2.80 (2.71)

19. Secondary Outcome: Positive and Negative Affect Scales - Positive Affect Scale (PANAS-Pos)
Description: Evaluation of positive affect collected at the end of each phase for male and female participants. Range 10 to 50, with higher scores indicating greater positive affect
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 83 | 76 | 81 | 71 | 74
Units on a scale | 32.30 (8.56) | 31.12 (9.25) | 32.82 (9.69) | 32.80 (9.40) | 31.65 (9.09) | 33.03 (8.76)

20. Secondary Outcome: Positive and Negative Affect Scales - Negative Affect Scale (PANAS-Neg)
Description: Evaluation of negative affect collected at the end of each phase for male and female participants. Range 10 to 50, with higher scores indicating greater negative affect
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 83 | 76 | 81 | 71 | 74
Units on a scale | 16.43 (7.31) | 16.22 (6.94) | 15.53 (6.89) | 17.19 (7.09) | 17.73 (8.06) | 16.07 (6.30)

21. Secondary Outcome: Smartphone Daily Measures of Nicotine Dependence Symptoms
Description: Evaluation of mean nicotine dependence symptoms collected daily during each phase. Range 1 to 5, with higher values indicating greater nicotine dependence symptoms
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 83 | 83 | 78 | 75 | 74 | 76
Units on a scale | 2.40 (0.35) | 2.42 (0.48) | 2.34 (0.42) | 2.44 (0.33) | 2.53 (0.37) | 2.42 (0.34)

22. Secondary Outcome: American Thoracic Society Questionnaire (ATSQ)
Description: Evaluation of respiratory symptoms collected at the end of each phase for male and female participants. Range 8 to 40, with higher numbers indicating more respiratory symptoms
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
Number analyzed (Participants) | 87 | 82 | 76 | 81 | 71 | 75
Units on a scale | 18.30 (8.98) | 16.85 (8.86) | 16.93 (8.59) | 18.17 (8.59) | 16.13 (7.96) | 16.08 (7.96)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Usual Brand Cigarette Phase (Men) | Placebo Standardized Research Electronic Cigarette Phase (Men) | Nicotine Standardized Research Electronic Cigarette Phase (Men) | Usual Brand Cigarette Phase (Women) | Placebo Standardized Research Electronic Cigarette Phase (Women) | Nicotine Standardized Research Electronic Cigarette Phase (Women)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/87 | 0/87 | 0/82 | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/87 | 1/87 | 3/87 | 1/82 | 1/82 | 2/82
Other Adverse Events (participants affected / at risk) | 0/87 | 0/87 | 0/87 | 0/82 | 0/82 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Brand Cigarette Phase (Men) (N=87) | Placebo Standardized Research Electronic Cigarette Phase (Men) (N=87) | Nicotine Standardized Research Electronic Cigarette Phase (Men) (N=87) | Usual Brand Cigarette Phase (Women) (N=82) | Placebo Standardized Research Electronic Cigarette Phase (Women) (N=82) | Nicotine Standardized Research Electronic Cigarette Phase (Women) (N=82)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flu Like Symptoms (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Psychosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03856515/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT03856515/ICF_001.pdf